CLINICAL TRIAL: NCT01570881
Title: Association of Plasma Melatonin Levels With Delirium After Sevoflurane Anesthesia
Brief Title: Association of Plasma Melatonin Levels With Delirium
Status: Completed | Type: Observational
Sponsor: Okayama University (Other)
Responsible Party: Principal Investigator, Shiho Yoshitaka, M.D., Okayama University
Other Study IDs: Okamasui3130
Record Dates: First submitted 2012-03-24; First posted 2012-04-04 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-04

CONDITIONS: Postoperative Delirium
Keywords: postoperative delirium; melatonin; sevoflurane
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Delirium,Nondelirium: those with delirium and those without delirium

SUMMARY:
Delirium is common complications in postoperative critically ill patients. However the mechanism of postoperative delirium is not well understood.The investigators designed a prospective observational study to investigate the association of perioperative plasma melatonin levels with postoperative delirium and general anesthesia. The investigators included 33 patients required intensive care more than 48 hours after sevoflurane anesthesia in an academic tertiary care hospital. The investigators measured plasma melatonin levels 4 times and assessed postoperative delirium using Confusion Assessment Method for the intensive care unit (CAM-ICU).

DETAILED DESCRIPTION:
Delirium is common complications in postoperative critically ill patients. Although the mechanism of postoperative delirium is not well understood, there are several studies to report alternation of plasma melatonin levels after general anesthesia and suggest the link between delirium and abnormal tryptophan-serotonin-melatonin metabolism. However, there are few studies to assess the association of perioperative plasma melatonin levels with postoperative delirium and/or general anesthetics.

The investigators designed a prospective observational study to investigate the association of perioperative plasma melatonin levels with postoperative delirium and general anesthesia. The investigators included 33 patients required intensive care more than 48 hours after sevoflurane anesthesia in an academic tertiary care hospital. The investigators measured plasma melatonin levels and assessed postoperative delirium using Confusion Assessment Method for the intensive care unit (CAM-ICU). The investigators compared perioperative plasma melatonin levels between patients with and without delirium, and assessed associations of patients' demographics and anesthesia with plasma melatonin levels.

ELIGIBILITY:
Inclusion Criteria:

* patients over 20 years of age who had undergone elective surgery with sevoflurane anesthesia and were expected to require postoperative intensive care for more than 48 hours

Exclusion Criteria:

* emergency surgery, history of psychosis and drug/alcohol abuse, and vision or hearing impairment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Okayama University Hospital with 22 beds in ICU.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2010-04; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The diagnose of postoperative delirium | One trained physician performed assessments of delirium at 1 hour after operation, and 8 AM and 5 PM of postoperative day 1 and 2.
  One trained physician performed assessments of delirium using Confusion Assessment Method for the intensive care unit at 1 hour after operation, and 8 AM and 5 PM of postoperative day 1 and 2.

SECONDARY OUTCOMES:
The measurements of plasma melatonin levels | We collected blood samples for the measurement of plasma melatonin levels at 1) 8 AM before operation, 2) 1 hour after operation, 3) 8 AM of postoperative day 1 and 4) 8 AM of postoperative day 2.
  We collected blood samples for the measurement of plasma melatonin levels at 1) 8 AM before operation, 2) 1 hour after operation, 3) 8 AM of postoperative day 1 and 4) 8 AM of postoperative day 2.Plasma was separated by centrifugation and the plasma was stored at least -30 degrees Celsius in a polypropylene tube until the time of assay. Plasma melatonin levels were measured with a melatonin radioimmunoassay kit (Buhlmann Laboratories AG, Allschwil, Switzerland).

CONTACTS AND LOCATIONS:
Overall Officials: Moritoki Egi, Principal Investigator — Department of Anesthesiology and Resuscitology, Okayama University
Locations (1):
- Okayama University, Okayama, Okayama-ken, Japan

REFERENCES:
- [Derived] Yoshitaka S, Egi M, Morimatsu H, Kanazawa T, Toda Y, Morita K. Perioperative plasma melatonin concentration in postoperative critically ill patients: its association with delirium. J Crit Care. 2013 Jun;28(3):236-42. doi: 10.1016/j.jcrc.2012.11.004. Epub 2013 Jan 9. PMID 23312124